CLINICAL TRIAL: NCT01262014
Title: Phase II, Multicenter, Prospective, Single Arm, Open Labeled Clinical Trial Investigating Pazopanib, a Multi-targeted Tyrosine Kinase Inhibitor (TKI) of VEGFR-1, -2, -3, PDGFR-α and -β and c-Kit in Patients With Platinum-resistant Advanced Ovarian Cancer.
Brief Title: Clinical Trial Investigating Pazopanib in Patients With Platinum-resistant Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICO-1002; 2010-020439-38 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Platinum-resistant Advanced Ovarian Cancer
Keywords: platinum; resistant; advanced; ovarian; cancer
MeSH Terms: conditions — Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental single arm (Experimental): Single arm of pazopanib 800 mg (2x400mg) given as a single agent.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg (2x400mg) pazopanib per day should be taken orally without food at least one hour before or two hours after a meal until disease progression, the development of unacceptable toxicity, noncompliance, withdrawal of consent by the patient, or investigator decision.

SUMMARY:
Given the low Responses Rates and short survival times achieved with conventional cytotoxic agents in resistant ovarian cancer patients, new treatment options are needed in this patient population.Antiangiogenic therapy has an important role in this group of patients and Pazopanib in particular. We are going to study if Pazopanib is able to control disease-related symptoms minimizing the side effects of treatment. This aspect is very important in the treatment of resistant ovarian cancer patient since our treatment is palliative without any impact in overall survival. So our goal is to study the Clinical Benefit Rate (objective responses plus stable disease rates) achieved with Pazopanib and its toxicity profile in this subgroup of patients

DETAILED DESCRIPTION:
Ovarian cancer is considered a chemo-responsive neoplasm, with initial response rates to systemic chemotherapy exceeding 80% when integrated with primary cytoreductive surgery Despite this, over 50% of women diagnosed with epithelial ovarian cancer eventually go on to die from their disease. Six major trials published over the past 15 years report that the median PFS for patients with advanced disease ranges between 16 and 23 months while the median OS lies between 31 and 65 months.The majority of patients who achieve a Complete Response with first-line chemotherapy ultimately develop recurrent disease. These patients can be subdivided into platinum-sensitive or platinum-resistant groups. In platinum-sensitive patients, disease recurrence occurs more than 6 months after cessation of initial platinum-containing chemotherapy. Platinum-based therapies are typically used to retreat these patients, in light of clinically meaningful responses observed in these patients following a second platinum-based treatment.Currently, there is no optimal treatment strategy for platinum-resistant patients whose disease recurs within 6 months of completing initial platinum-based chemotherapy.Despite a wide range of available treatments, prolonged survival has not been shown in this setting, and ORR is generally less than 20%. As resistant-disease is not curable, the goals of treatment for these patients include palliation of symptoms and improvements in quality of life. Platinum-resistance is therefore a significant clinical problem for which improved treatment regimens are needed. In this regard, molecular targeted therapeutic agents herald a new era for cancer treatment. In the setting of epithelial ovarian cancer, a growing body of evidence supports the use of anti-angiogenic agents.Platinum-resistant ovarian cancer patients are often treated with sequential lines of single-agent chemotherapy. Commonly used agents include topotecan, pegylated liposomal doxorubicin (PLD), weekly paclitaxel and gemcitabine.Topotecan is topoisomerase I inhibitor well established as therapy for recurrent ovarian cancer, with demonstrated efficacy in platinum-resistant populations. PLD is licensed in the US and Europe for use in ovarian cancer after failure of platinum chemotherapy and is recommended by the NCCN as a treatment option in this setting. PLD and topotecan have been compared in a Phase III study of 474 patients with tumours that were recurrent or refractory to platinum-based chemotherapy. In the subgroup of patients with platinum-resistant tumours treated with PLD (n=130), the ORR was 12.3%, and median PFS and OS were 2.1 and 8.2 months, respectively. The 124 platinum-resistant patients who received topotecan achieved median PFS and OS of 3.1 months and 9.5 months, respectively, which were not significantly different from the PLD group. For platinum-resistant patients, outcomes were not significantly different between treatment groups so whatever treatment option is acceptable.In a recent study in platinum-resistant recurrent ovarian cancer patients, topotecan monotherapy showed and ORR of 19% and 9% when used as conventional or weekly schedule, respectively. Angiogenesis is known to play a critical role in the growth of ovarian tumours and may represent an important target. For example, several studies have demonstrated that increased microvessel density in primary ovarian tumours is associated with VEGF expression and predicted worsened survival rates. Likewise, circulating VEGF levels were significantly higher in ovarian cancer subjects with an advanced stage at diagnosis, poorly-differentiated tumours, or increased levels of ascites as compared to subjects with an early stage, well-differentiated tumour(s), and less ascites. Tumour-derived VEGF may play a role in ascites formation. Angiogenesis has been shown to be a negative predictive factor for overall survival and disease-free survival in women with advanced ovarian cancer 18. Blockade or inhibition of VEGF (eg, using bevacizumab) or VEGFR (using TKIs) have been shown to be effective in Phase II studies in ovarian cancer. For example, single-agent bevacizumab has shown a 16-21% overall tumour response rate (ORR) in two studies of previously treated patients with ovarian cancer.Pazopanib is a potent, multi-targeted tyrosine kinase inhibitor (TKI) of VEGFR-1, -2, -3, PDGFR-α and -β and c-Kit. Pazopanib has shown evidence of antitumor activity in clinical studies of ovarian cancer. VEG104450 is a Phase II study of pazopanib in subjects with ovarian, fallopian tube, or primary peritoneal cancers who had responded to first-line chemotherapy and who were at high risk of clinical recurrence (as evidenced by rising CA-125 levels). 36 subjects were enrolled, of which 22 (61%) had a sensitive platinum relapse and a previous chemotherapy regimen. Final results obtained recently indicate the following:10 out of 36 (28%) subjects experienced a CA-125 response to pazopanib with responses occurring shortly after start of pazopanib administration (median time to response 29 days) with a median duration of response of 113 days 21.Taking into account theses results, pazopanib is one of the promising antiangiogenic therapies to be studied against ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.
2. Age ≥ 18 years
3. The patient has histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. The patient has completed at least 4 CYCLES OF one and up to two platinum-containing regimens (involving cisplatin or carboplatin),for the management of this condition. Treatment may have included intraperitoneal therapy, consolidation or extended therapy administered after surgical or nonsurgical assessment.
6. The patient must have a platinum-free interval of ≤ 6 months after the final dose of primary or subsequent platinum-based therapy.

   Patients must have platinum-resistant disease,(defined as progression within <6 months from completion of a minimum of 4 platinum therapy cycles. The date should be calculated from the last administered dose of platinum therapy.
7. The patient has at least one unidimensionally measurable target lesion (≥ 20 mm or ≥ 10 mm by spiral computed tomography [CT] or magnetic resonance imaging [MRI]), as defined by Response Evaluation Criteria in Solid Tumors (RECIST) guidelines V 1.1.
8. Previously archived tumor tissue from either the primary or metastatic tumor (paraffin block or 10 unstained slides) should be collected prior to administration of the first dose of study therapy and stored at a secure central laboratory.
9. Adequate organ system function
10. Women of child bearing potential should be using an effective method of contraception (complete abstinence, any intrauterine device (IUD) with published data showing that the lowest expected failure rate is < 1 % per year; or any other methods with published data showing that the lowest expected failure rate is less than 1 % per year) before entry into the study and throughout the same and for 6 months after ending the study. Women of childbearing potential must have a negative test serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta human chorionic gonadotropin [β-HCG]) within 7 days prior to randomization.
11. Able to swallow oral compound.
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

1. Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
2. Previous treatment with >2 anticancer regimens for ovarian cancer
3. Prior treatment with any antiangiogenic treatment (i.e. Bevacizumab)
4. Patients with platinum-refractory disease defined as those patients progress during platinum-based therapy.
5. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
6. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.

     * active episodes of intestinal pseudo-obstruction
7. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   * Malabsorption syndrome
   * Major resection of the stomach or small bowel.
   * Grade 3 diarrhoea
8. Presence of uncontrolled infection.
9. Corrected QT interval (QTc) > 480 msecs using Bazett's formula
10. History of any one or more of the following cardiovascular conditions within the past 6 months:

    * Cardiac angioplasty or stenting
    * Myocardial infarction
    * Unstable angina
    * Coronary artery bypass graft surgery
    * Symptomatic peripheral vascular disease
    * Class II, III or IV congestive heart failure, as defined by the New York Heart Association (NYHA
11. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg] instead an anti-hypertensive treatment.

    Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be assessed using the following recommendations:

    Once a patient has had an elevated blood pressure reading (> 140/80mmHg) this should be confirmed with another measurement, done locally if possible, either by the patients local doctor, or by home monitoring if available. Patients should continue to have their blood pressure monitored, at least weekly, until it becomes controlled (i.e. ≤ 140/80mmHg on 2 separate occasions, at least one week apart). Anti-hypertension medication changes, such as initiation of therapy, dose increases of existing therapies, or addition of other anti-hypertensive agents, should be done if the blood pressure remains high at 2 consecutive readings, at least 24 hours apart. Please, refer to guidance regarding the management of hypertension for the patient's local doctor for further information.
12. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

    Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
13. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
14. Prior minor surgery within 7 days prior to first dose of study drug
15. Evidence of active bleeding or bleeding diathesis.
16. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
17. Hemoptysis within 6 weeks of first dose of study drug.
18. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
19. Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
20. Treatment with any of the following anti-cancer therapies:

    radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
21. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
22. Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint for this study is Clinical Benefit Rate | average 30 months
  Clinical Benefit Rate defined as the percentage of patients with Complete Response plus Partial Response plus Stable Disease ≥ 8 weeks by RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | average 30 months
  Progression Free Survival (PFS) is defined as the time from the day of starting treatment to the first evidence of progression as defined by RECIST guidelines (v1.1) or death from any cause. If the patient does not have a documented date of progression or death, then PFS will be censored at the date of last adequate assessment.
Biological Response by CA-125 (GCIG Criteria) | average 30 months
  CA-125 Testing: at pretreatment visit and during the treatment period and then every 3 months after discontinuation of treatment due to any reason (toxicity or patient will) until disease progression.
Overall Survival (OS) | Average 3 years
  Overall Survival (OS) is defined as the time from first day of therapy to the date of death from any cause. For a patient who is alive at the time of the statistical analysis, the patient will be considered censored at the last date of known contact.
Biological progression-free interval (PFIBIO) | average 30 months
  CA-125 Testing: at pretreatment visit and during the treatment period and then every 3 months after discontinuation of treatment due to any reason (toxicity or patient will) until disease progression. PFIBIO will be assessed according to the GCIG criteria
Quality of Life and symptom control | average 5 years
  Quality of Life and symptom control will be assessed using EORTC QLQ-C30, QLQOV28, FACT/NCCN Ovarian Symptom Index (FOSI)
The safety and tolerability of study drug | Average 5 years
  The safety and tolerability of study drugs are determined type, incidence, severity, timing, seriousness, and relatedness; of reported AEs, physical examinations, and laboratory tests. Toxicity will be graded and tabulated by the NCI-CTCAE v 3.0.
Descriptive pharmacodynamic profile | 30 months
  * the association between tumor PDGFRα expression (assessed by immunohistochemistry) and clinical outcomes (PFS, ORR, etc)
  * the relationship between serum VEGF/PDGF levels and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, MD, Study Chair — H Vall d'Hebron
Locations (20):
- Spain (20):
  - H. Alcorcón, Alcorcón
  - H. de la Santa Creu i Sant Pau, Barcelona
  - H Vall d'Hebron, Barcelona
  - H. Clínic Barcelona, Barcelona
  - H Reina Sofía Cordoba, Córdoba
  - Intitut Català d' Oncolgia L' Hospitalet, L'Hospitalet de Llobregat
  - HGU Gregorio Marañón, Madrid
  - Centro Oncológico MD Anderson Spain, Madrid
  - H Ramón y Cajal de Madrid, Madrid
  - H Madrid. Centro Integral Oncológico Clara Campal, Madrid
  - H de Sant Joan de Deu, Manresa
  - H Morales Meseguer, Murcia
  - H Son Dureta, Palma de Mallorca
  - H Son Llatzer, Palma de Mallorca
  - H. Parc Taulí, Sabadell
  - H Marqués de Valdecilla, Santander
  - H La Fe de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - H General de Valencia, Valencia
  - H Miguel Servet, Zaragoza